CLINICAL TRIAL: NCT04378868
Title: Role of Delay and Antibiotics on PERForation Rate While Waiting appendECTomy - Randomized Non-inferiority Trial
Brief Title: Role of Delay and Antibiotics on Perforation Rate While Waiting Appendectomy
Acronym: PERFECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Panu Mentula, Adjunct Professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS-PERFECT; 2019-002348-26 (EudraCT Number)
Record Dates: First submitted 2020-04-29; First posted 2020-05-07 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Anti-Bacterial Agents; Cefuroxime; Metronidazole

STUDY DESIGN:
Intervention Model Description: Patients are randomized into two arms according to urgency and simultaneously each patient is randomized into two arms according to antibiotic treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Surgery within 8 hours, no antibiotics (Active Comparator): Patients are planned for urgent operation, that should be done within 8 hours. Operation can be done during the night time. Patients do not receive antibiotics while waiting surgery. Prophylactic antibiotics are given 0-30 minutes before incision.
  Interventions: Drug: No antibiotics; Other: urgent schedule
- Surgery within 24 hours, no antibiotics (Experimental): Patients are planned for urgent operation, that should be done within 24 hours. Operations are not done during the night time (00:00 - 08:00), unless necessary to avoid delay over 24 hours. Patients do not receive antibiotics while waiting surgery. Prophylactic antibiotics are given 0-30 minutes before incision.
  Interventions: Drug: No antibiotics; Other: less urgent schedule
- Surgery within 8 hours, antibiotics (Experimental): Patients are planned for urgent operation, that should be done within 8 hours. Antibiotics (cefuroxime 1.5g and metronidazole 500mg every 8 hours) are given while waiting surgery.
  Interventions: Drug: Antibiotics, cefuroxime and metronidazole; Other: urgent schedule
- Surgery within 24 hours, antibiotics (Experimental): Patients are planned for urgent operation, that should be done within 24 hours. Operations are not done during the night time (00:00 - 08:00), unless necessary to avoid delay over 24 hours. Antibiotics (cefuroxime 1.5g and metronidazole 500mg every 8 hours) are given while waiting surgery.
  Interventions: Drug: Antibiotics, cefuroxime and metronidazole; Other: less urgent schedule

INTERVENTIONS:
Drug: Antibiotics, cefuroxime and metronidazole — Patient receives antibiotics while waiting appendectomy
  Arms: Surgery within 24 hours, antibiotics; Surgery within 8 hours, antibiotics
Drug: No antibiotics — No antibiotics are given while waiting surgery.
  Arms: Surgery within 24 hours, no antibiotics; Surgery within 8 hours, no antibiotics
Other: urgent schedule — Patients can wait up to 8 hours for surgery.
  Arms: Surgery within 8 hours, antibiotics; Surgery within 8 hours, no antibiotics
Other: less urgent schedule — Patients can wait up to 24 hours for surgery.
  Arms: Surgery within 24 hours, antibiotics; Surgery within 24 hours, no antibiotics

SUMMARY:
This study evaluates the effects of preoperative delay and antibiotics on perforation rate of appendix while waiting surgery for acute appendicitis. Patients with diagnosed acute appendicitis are randomized into two urgency groups: surgery within 8 hours or surgery within 24 hours. In addition, patients are randomized to either receive antibiotics while waiting or waiting without antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Acute appendicitis where surgery is planned. Diagnosis of appendicitis should be verified either by clinical diagnosis with Adult Appendicitis Score >=16 or by diagnostic imaging (CT-scan, MRI or ultrasound) showing appendicitis. All patients with symptoms at least 3 days should undergo diagnostic imaging before inclusion.

Exclusion Criteria:

* Complicated appendicitis according to diagnostic imaging. The following findings indicate complicated appendicitis: extraluminal air or extraluminal fecalith; fluid collection, abscess or phlegmon next to appendix; non-enhancement appendiceal wall on contrast enhanced CT-scan.
* Plasma C-reactive protein >=100
* Fever measured on emergency department over 38.5 degrees Celcius.
* Clinical generalized peritonitis or other reason that indicate immediate surgery
* Pregnancy, pregnancy test is taken from all fertile aged women before randomization
* Allergy to study antibiotics, or anaphylactic reaction after betalactam antibiotic or other contraindication for metronidazole or ongoing antibiotic treatment or patient is carrier of resistant bacteria. (This exclusion criteria are applicable only on randomization into antibiotic treatment arms)
* Missing written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Complicated appendicitis | during surgery
  Surgical finding is complicated appendicitis (AAST Grade III-V)

SECONDARY OUTCOMES:
Time of hospital stay | 30 days from surgery
  Time in hours from randomization to discharge from hospital
Postoperative complications | 30 days from surgery
  complications are defined according to Clavien-Dindo classification
Pain measured by numeric rating scale while waiting surgery | up to 36 hours
  Pain is measured by numeric rating scale (NRS) every hour by patient, and area under NRS represents overall pain.
Surgical site infections (SSI) and positive blood cultures | within 30 days from randomization
  SSIs classified according to CDC classification: superficial incisional, deep incisional and organ/space infection. Blood cultures are obtained if patient has fever over 38.5 degrees Celcius.
Conversions of laparoscopic surgeries to open surgery | during the the first operation for acute appendicitis
  All surgeries are started as laparoscopic surgery. Conversion means that operation is converted to open surgery during the same operation.
Gangrenous or perforated appendicitis according to pathological examination. | 3 week after surgery
  All specimens are sent to pathological examination and all pathological reports are reviewed
Sunshine Appendicitis Grading System Score classification | during surgery
  Sunshine Appendicitis Grading System Score (range 0-4) for appendicitis. Higher score represents worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Panu J Mentula, MD, Principal Investigator — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - HUS, Jorvi Hospital, Espoo
  - HUS, Meilahti Hospital, Helsinki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sammalkorpi HE, Mentula P, Leppaniemi A. A new adult appendicitis score improves diagnostic accuracy of acute appendicitis--a prospective study. BMC Gastroenterol. 2014 Jun 26;14:114. doi: 10.1186/1471-230X-14-114. PMID 24970111
- [Background] Shafi S, Aboutanos M, Brown CV, Ciesla D, Cohen MJ, Crandall ML, Inaba K, Miller PR, Mowery NT; American Association for the Surgery of Trauma Committee on Patient Assessment and Outcomes. Measuring anatomic severity of disease in emergency general surgery. J Trauma Acute Care Surg. 2014 Mar;76(3):884-7. doi: 10.1097/TA.0b013e3182aafdba. PMID 24553565
- [Background] Reid F, Choi J, Williams M, Chan S. Prospective evaluation of the Sunshine Appendicitis Grading System score. ANZ J Surg. 2017 May;87(5):368-371. doi: 10.1111/ans.13271. Epub 2015 Sep 1. PMID 26333132
- [Derived] Jalava K, Sallinen V, Lampela H, Malmi H, Steinholt I, Augestad KM, Leppaniemi A, Mentula P. Role of preoperative in-hospital delay on appendiceal perforation while awaiting appendicectomy (PERFECT): a Nordic, pragmatic, open-label, multicentre, non-inferiority, randomised controlled trial. Lancet. 2023 Oct 28;402(10412):1552-1561. doi: 10.1016/S0140-6736(23)01311-9. Epub 2023 Sep 14. PMID 37717589
- [Derived] Jalava K, Sallinen V, Lampela H, Malmi H, Leppaniemi A, Mentula P. Role of delay and antibiotics on PERForation rate while waiting appendicECTomy (PERFECT): a protocol for a randomized non-inferiority trial. BJS Open. 2021 Sep 6;5(5):zrab089. doi: 10.1093/bjsopen/zrab089. PMID 34580704
- See also: Link for calculation of Adult Appendicitis Score — https://www.appendicitisscore.com